CLINICAL TRIAL: NCT00509561
Title: A Randomised Phase II/III Multi-Centre Clinical Trial of Definitive Chemotherapy, With or Without Cetuximab, in Carcinoma of the Oesophagus
Brief Title: Cisplatin, Capecitabine, and Radiation Therapy With or Without Cetuximab in Treating Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wales Cancer Trials Unit (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000558804; WCTU-SCOPE-1; EU-20739; EUDRACT-2006-002241-37; ISRCTN47718479; CTA-17853/0202/001-0001
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage IA esophageal cancer; stage IB esophageal cancer; stage IIA esophageal cancer; stage IIB esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cetuximab; Capecitabine; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemo-radiotherapy (Active Comparator)
  Interventions: Drug: capecitabine; Drug: cisplatin; Radiation: radiation therapy
- Chemo-radiotherapy plus cetuximab (Experimental)
  Interventions: Biological: cetuximab; Drug: capecitabine; Drug: cisplatin; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab
  Arms: Chemo-radiotherapy plus cetuximab
Drug: capecitabine
Drug: cisplatin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and capecitabine, work in different ways to kill tumor cells or stop them from growing. Radiation therapy uses high-energy x-rays to kill tumor cells. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving cisplatin together with capecitabine and radiation therapy is more effective with or without cetuximab in treating esophageal cancer.

PURPOSE: This randomized phase II/III trial is studying the side effects and how well giving cisplatin together with capecitabine, radiation therapy, and cetuximab works compared with giving cisplatin, capecitabine, and radiation therapy without cetuximab in treating patients with esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether the addition of cetuximab to definitive chemoradiotherapy comprising cisplatin, capecitabine, and radiotherapy shows evidence of enhanced overall survival in patients with carcinoma of the esophagus.
* To determine the safety of this regimen in these patients.
* To determine the feasibility of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cisplatin IV over 2 hours on days 1, 22, 43, and 64 and oral capecitabine twice daily on days 1-84. Beginning in week 7 patients also undergo radiotherapy 5 days a week for 5 weeks (weeks 7-11). Treatment continues in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive cisplatin and capecitabine and undergo radiotherapy as in arm I. Patients also receive cetuximab IV over 1-2 hours on day 1 in weeks 1-12. Treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life and health economics are assessed at baseline, during treatment, and at pre-specified time points during follow-up.

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for 1 year, and then annually for a minimum of 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the esophagus

  * Adenocarcinoma
  * Squamous cell
  * Undifferentiated carcinoma
  * Siewert type I tumor of the gastroesophageal junction
* Localized, nonmetastatic disease (T1-4, N0-1) confirmed by endoscopic ultrasound (EUS) and spiral CT scan
* Total disease length (primary and lymph nodes) < 10 cm by EUS
* Not suitable for surgery (either for medical reasons or patient's choice)
* No metastatic disease (i.e., M1a or M1b according to UICC TNM version 6)
* No significant (> 2 cm) extension of tumor into the stomach

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* White blood cell count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL (should be corrected to > 10 g/dL before treatment)
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT/AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 3 times ULN
* Glomerular filtration rate > 40 mL/min OR > 60 mL/min estimated by Cockcroft-Gault formula
* Adequate cardiac ejection fraction ≥ 40% by MUGA or ECHO
* FEV_1 ≥ 1 L by spirometry
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No malignancy within the past 5 years
* No unstable angina, uncontrolled hypertension, cardiac failure, or other clinically significant cardiac disease
* No major trauma within the past 4 weeks
* No known dihydropyrimidine dehydrogenase deficiency
* No hearing impairment or sensory-motor neuropathy > grade 2

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior sorivudine and analogues
* At least 4 weeks since prior major surgery
* At least 4 weeks since prior monoclonal antibody
* At least 3 months since prior radiotherapy
* No prior treatment for invasive esophageal carcinoma or gastroesophageal junction carcinoma (not including photodynamic therapy or laser therapy for high-grade dysplasia/carcinoma in situ)
* No other prior treatment for this malignancy that would compromise the ability to deliver definitive mediastinal chemoradiotherapy or compromise survival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2008-02; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Treatment-failure rate at 24 weeks
Overall survival

SECONDARY OUTCOMES:
Feasibility
Toxicity
Quality of life
Quality of assurance
Health economics

CONTACTS AND LOCATIONS:
Overall Officials: Tom Crosby, MD, Study Chair — Velindre NHS Trust
Locations (55):
- United Kingdom (55):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Good Hope Hospital, Birmingham, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Cumberland Infirmary, Carlisle, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Gloucestershire Royal Hospital, Cheltenham, England
  - Walsgrave Hospital, Coventry, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Princess Alexandra Hospital, Essex, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Cookridge Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Lincoln County Hospital, Lincoln, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Helen Rollason Cancer Care Centre at North Middlesex Hospital, London, England
  - University College of London Hospitals, London, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital, Nottingham, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Derriford Hospital, Plymouth, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Alexandra Healthcare NHS, Redditch, England
  - Scarborough General Hospital, Scarborough, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Southampton General Hospital, Southampton, England
  - Southport and Formby District General Hospital, Southport, England
  - Royal Marsden - Surrey, Sutton, England
  - Musgrove Park Hospital, Taunton, England
  - Torbay Hospital, Torquay, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Worcester Royal Hospital, Worcester, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - Singleton Hospital, Swansea, Wales
  - Wrexham Maelor Hospital, Wrexham, Wales